CLINICAL TRIAL: NCT00638937
Title: A Phase 2 Study of AZD0530 in Patients With Advanced, Recurrent Non-Small Cell Lung Cancer Who Have Previously Received Platinum-Based Combination Chemotherapy
Brief Title: AZD0530 to Treat Recurrent Stage IIIB/IV NSCLC Previously Treated With Combination Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01053; NCI-2009-01053 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PMH-PHLO-053 (Other Grant/Funding Number: N01CM00032); CDR0000587610 (Other Grant/Funding Number: N01CM00032); PHL-053 (Other: University Health Network-Princess Margaret Hospital); 7555 (Other: CTEP); N01CM00032 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2008-03-18; First posted 2008-03-19 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (saracatinib) (Experimental): Patients receive saracatinib PO, at a dose of 175 mg QD on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib — Given PO
  Other Names: AZD0530

SUMMARY:
This phase II trial is studying how well saracatinib works in treating patients with recurrent, stage IIIB or stage IV non-small cell lung cancer previously treated with combination chemotherapy that included cisplatin or carboplatin. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the rate of disease control (i.e., lack of disease progression, a combined rate of objective complete and partial response, and stable disease) for at least 4 cycles of therapy in patients with AZD0530 (saracatinib) in patients with advanced non-small cell lung cancer that had previously been treated with platinum-based combination chemotherapy.

SECONDARY OBJECTIVES:

I. To assess the objective response rate (complete and partial response), stable disease rate, duration of response or stable disease, progression-free, median and 6 month overall survival rates, safety and tolerability of this treatment.

TERTIARY OBJECTIVES:

I. To evaluate potential predictive markers by assessing pretreatment intratumoral levels of src, Y419 phospho-src (P-Src) and c-terminal src kinase (Csk) in archival tumor biopsies.

OUTLINE: This is a multicenter study.

Patients receive saracatinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected at baseline and at 2 weeks after beginning treatment and are analyzed for c-Src protein expression and activity by immunofluorescence staining. P-glycoprotein levels and phosphorylation of focal adhesion kinase (FAK), paxillin, caveolin, and Stat-3 are also measured using tumor tissue samples. Blood samples are also used to measure levels of vascular endothelial growth factor (VEGF) by enzyme-linked immunosorbent assay (ELISA).

After completion of study treatment, patients are followed every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent/metastatic/locally advanced unresectable, histologically or cytologically confirmed NSCLC
* Measurable disease defined (RECIST) as at least 1 lesion measured in at least 1 dimension (longest diameter) as >20mm with conventional techniques or >10mm with spiral CT scan
* Previously treated with firstline platinum-based systemic chemotherapy for advanced disease AND had at least disease stabilization as best response to firstline therapy

  * <=1 line of prior therapy
  * Not have had prior treatment with EGFR Tyrosine kinase inhibitor
  * Completed chemotherapy/surgery/radiotherapy 4 weeks before study entry and must have recovered from toxic effects of prior therapy
  * Had >40% of their bone marrow radiated and must have either measurable disease outside field/documented progression post radiation therapy
* Life expectancy >3 months
* ECOG performance status =<2 OR Karnofsky >=60%
* Leukocytes >=3x10^9/L
* Absolute neutrophil count >=1.5x10^9/L
* Platelet count >=10x10^9/L
* Hemoglobin >9g/dL (may be transfused to meet this)
* Total bilirubin =<1.5 times institutional ULN (IULN)
* AST/ALT =<2.5xIULN (=<5 times ULN in the presence of liver metastases)
* Creatinine =<1.5xIULN OR creatinine clearance >=50 mL/min/1.73m^2
* Urine protein creatinine ratio =<1.0 OR urine protein >1.0, 24 hour urine for protein should be <1000mg
* Women of childbearing potential/men must use adequate contraception (hormonal/barrier method of birth control; abstinence) prior to study entry, for duration of study participation, and for 8 weeks following cessation of study therapy
* Ability to understand/willingness to sign written informed consent

Exclusion Criteria:

* Chemotherapy/radiotherapy within 4 weeks (6 weeks for nitrosoureas/mitomycin C) prior to study entry/not recovered from AEs due to agents administered > than 4 weeks earlier
* No CYP3A4-active agents permitted during protocol treatment. Patients requiring treatment with these agents are not eligible; prohibited drugs should be discontinued 7 days before first dose of AZD0530 and for 7 days after discontinuation of AZD0530
* Cannot receive other investigational agents
* History of allergic reactions attributed to compounds of similar chemical/biologic composition to AZD0530
* QTc prolongation (i.e.QTc interval >=460 msec)/other significant ECG abnormalities
* Poorly controlled hypertension (i.e.systolic BP of 140 mmHg or higher, diastolic BP of 90mm Hg or higher)
* Any condition impairing ability to swallow AZD0530 tablets
* Treated brain metastases which are clinically and radiologically stable are permitted; patients requiring steroids/with neurological symptoms should be excluded because of poor prognosis/often develop progressive neurologic dysfunction
* Intercurrent cardiac dysfunction including but not limited to symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia are excluded as are those with ischemic heart disease history including myocardial infarction
* Uncontrolled intercurrent illness including but not limited to ongoing/active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women excluded because AZD0530 has potential teratogenic/abortifacient effects; because unknown but potential risks for AEs in nursing infants secondary to treatment of mother with AZD0530, breastfeeding should be discontinued if mother is treated with AZD0530
* HIV-positive patients on combination antiretroviral therapy are ineligible because potential for PK interactions with AZD0530; these patients have increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Laurie, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre (Ottawa Health Research Institute) Civic Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Saracatinib): Patients receive saracatinib PO QD on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression
  saracatinib: 175mg given PO daily
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Saracatinib)
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Saracatinib): Patients receive saracatinib PO QD on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression
  saracatinib: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 65 [33 to 78]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 37

OUTCOME MEASURES:

1. Primary Outcome: Rate of Disease Control (Freedom From Disease Progression)
Description: Lack of disease progression, a combined rate of objective complete (disapprearance of all target lesions) and partial responses (>= 30% decrease in sum of longest diameter of target lesions) and stable disease as determined by Response Evaluation Criteria in Solid Tumours (RECIST 1.0) for at least 4 cycles (16 weeks) of therapy.
  Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: 112 days
Measure: Number; unit: participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
participants | 4

2. Secondary Outcome: Objective Response Rate (Complete and Partial Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions Overall Response (OR) = CR + PR
  Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: From the start of the treatment until the criteria for response are met
Measure: Number; unit: participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
participants | 2

3. Secondary Outcome: Stable Disease Rate
Description: Stabilization of disease for atleast 4 cycles, leading to disease control
  Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: From the start of the treatment until the criteria for progression are met, assessed up to 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
participants | 4

4. Secondary Outcome: Duration of Response or Stable Disease
Description: Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: From first response until the criteria for progression are met, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
months | 1.8 [1.6 to 2.8]

5. Secondary Outcome: Median Progression-free Survival
Description: The Kaplan-Meier method will be used.
Time Frame: From the date of study enrollment to the time the criteria for disease progression are met, death or last contact, or the last tumor assessment before the initiation of further anticancer therapy, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 31
months | 1.8 [1.6 to 2.8]

6. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from randomization to the date of first documented disease progression or death from any cause
  The Kaplan-Meier method will be used.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
months | 1.8 [1.6 to 2.8]

7. Secondary Outcome: Median Overall Survival
Description: The Kaplan-Meier method will be used.
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
months | 7.6 [5.2 to 17.1]

8. Secondary Outcome: Overall Survival
Description: One year overall survival rate
  The Kaplan-Meier method will be used.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 37
percentage of participants | 43

ADVERSE EVENTS:
Arm/Group | Treatment (Saracatinib)
Serious Adverse Events (participants affected / at risk) | 10/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Saracatinib) (N=37)
Death NOS (General disorders) | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
INR increased (Investigations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic event (Vascular disorders) | 2
Fever (General disorders) | 2
Lung infection (Infections and infestations) | 1
Carbon monoxide diffusing capacity decreased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Saracatinib) (N=37)
Carbon monoxide diffusing capacity decreased (Investigations) | 33
Forced expiratory volume decreased (Investigations) | 33
Anemia (Blood and lymphatic system disorders) | 29
Fatigue (General disorders) | 29
Vital capacity abnormal (Investigations) | 28
Anorexia (Metabolism and nutrition disorders) | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24
Lymphocyte count decreased (Investigations) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less